CLINICAL TRIAL: NCT04104074
Title: A Pilot Study to Evaluate the Safety and Efficacy of Radiotherapy Plus Sintilimab for Advanced Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis
Brief Title: Safety and Efficacy of Radiotherapy Plus Sintilimab for HCC With Portal Vein Tumor Thrombosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19048-0-01
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Hepatocellular Carcinoma; Portal Vein Tumor Thrombosis
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiotherapy; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy Plus Sintilimab (Experimental): HCC Patients will be received radiotherapy and concurrent Sintilimab (PD-1 inhibitor)treatment.
  Interventions: Radiation: Radiotherapy; Drug: Sintilimab

INTERVENTIONS:
Radiation: Radiotherapy — Arm 1: The single radiotherapy dose was 200cGy, once a day, and the total dose was 5000cGy.
  Arm 2: the single dose of radiotherapy was 300 cGy, once a day, and the total dose was 3000 cGy.
Drug: Sintilimab — Sintilimab is a PD-1 inhibitor, intravenously, at a dose of 200 mg, once every 3 weeks
  Other Names: IBI308

SUMMARY:
The proposed study is an open-label, single-center, single arm phase 1b study to evaluate the safety and efficacy of radiotherapy plus sintilimab for HCC with PVTT.

DETAILED DESCRIPTION:
The patients were divided into two groups. The first group: the single dose of radiotherapy was 200 cGy, once a day, the total dose was 5000 cGy. The second group: the single dose of radiotherapy was 300 cGy, once a day, and the total dose was 3000 cGy.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent document.
2. Locally advanced hepatocellular carcinoma with identified tumor thrombosis of main portal vein or primary branches (left and / or right branches)
3. Has at least 1 measurable lesion
4. Age ≥18 years
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
6. Adequate organ function
7. Child Pugh class A
8. Life expectancy ≥12 weeks.
9. Antiviral therapy per local standard of care for hepatitis B
10. Woman of child bearing potential must have a negative pregnancy test
11. Must use acceptable form of birth control while on study

Exclusion Criteria:

1. Has previously been performed by raditotherapy for the area to be treated.
2. With extrahepatic metastasis
3. History of hepatic encephalopathy or liver transplantation
4. Untreated hepatitis infection: HBV DNA>2000IU/mlor10000 copy/ml, HCV RNA> 1000copy/ml, both HbsAg and anti-HCV body are positive
5. Has liver tumor not amenable to radiotherapy, or has had prior upper abdominal radiation therapy within planned volumes
6. Has had esophageal or gastric variceal bleeding within 3 months prior to study enrollment
7. With serious systemic diseases such as heart disease and cerebrovascular disease, and the condition is unstable or uncontrollable
8. Evidence of active pulmonary tuberculosis (TB)
9. Positive test of immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)
10. History of allergic reactions to related drugs

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 1 year
  Safety and tolerability of radiotherapy plus sintilimab based on NCI CTCAE v4.03 and RTOG/EORTC criteria

SECONDARY OUTCOMES:
Overall response rate (ORR) | 1 year
  Objective response rate based on RECIST v1.1 criteria
Progression-free survival (PFS) | 2 years
Overall Survival (OS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gong Li, MD, Principal Investigator — Beijing Tsinghua Changgeng Hospital
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality, China